CLINICAL TRIAL: NCT06893679
Title: Effects of Qigong Sensory Training on Sensory Modulation and Behavior in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR/AHS/24/0738
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Autism
Keywords: Qigong sensory training; Autism; Sensory Modulation; Strength; Behavior
MeSH Terms: conditions — Autistic Disorder; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Qigong sensory training (Experimental): Participants will be received 15 mints massage therapy 2 times in a day and 5 days a week for 8 weeks. Before and after 8 week of intervention, Assessment of sensory modulation scale (ASMS) will be used to check the sensory modulation level and strength and difficulties questionnaire (SDQ) will be used to check the behavior. Data will be collected from Nishtar Hospital Multan. The pre and post intervention assessments will be done.
  Interventions: Other: Qigong sensory training

INTERVENTIONS:
Other: Qigong sensory training — Participants will be received 15 mints massage therapy 2 times in a day and 5 days a week for 8 weeks. Before and after 8 week of intervention, Assessment of sensory modulation scale (ASMS) will be used to check the sensory modulation level and strength and difficulties questionnaire (SDQ) will be used to check the behavior. Data will be collected from Nishtar Hospital Multan. The pre and post intervention assessments will be done.

SUMMARY:
Autism Spectrum Disorder (ASD) is a complex neurodevelopmental condition characterized by challenges in social interaction, communication, and a range of repetitive behaviors. Among these challenges, sensory processing abnormalities are highly prevalent, manifesting as hyper- or hypo-sensitivity to sensory stimuli, and can significantly impact daily functioning and quality of life. In sensory modulation there are difficulties in regulating and responding appropriately to sensory input from the environment. Sensory modulation can have a significant impact on the daily lives of individuals with autism, affecting their ability to engage in various activities and navigate social interactions. Autistic children also have repetitive behaviors, such as repetitive actions like self-stimulation behavior, or stimming. These behaviors can involve one part of the body, the entire body or an object. QST in which deep pressure with thumb apply on head, neck, trunk and limbs along deep breathing which give relaxation to body and have effect on sensory modulation and behavior in children with Autism. The intended project aims to evaluate the sensory modulation and behavior in children with autism spectrum disorder (ASD) through Qigong Sensory Training (QST).

A quasi-Experimental study will be conduct to evaluate the effect of QST on the sensory modulation and behavior of autistic children. 21 Participants will be included in the study with age of 4-12 years diagnosed with ASD. Participants will be received 15 mints massage therapy 2 times in a day and 5 days a week for 8 weeks. Before and after 8 week of intervention, Assessment of sensory modulation scale (ASMS) will be used to check the sensory modulation level and strength and difficulties questionnaire (SDQ) will be used to check the behavior. Data will be collected from Nishtar Hospital Multan. The pre and post intervention assessments will be done. The reliability and validity of tools are mentioned. The duration of study will be 10-months. Data will be analyzed with the help of SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to12 years diagnosed with autism spectrum disorder.
* Male and Female will be included in study.
* Parental/guardian consent to participate in the study.
* Children do not receive any other intervention therapy during study

Exclusion Criteria:

* Children with severe physical disabilities that significantly impair their ability to participate in touch-based interventions, as determined by a qualified healthcare provider.
* Children diagnosed with severe psychiatric conditions other than autism spectrum disorder (ASD), including but not limited to schizophrenia, bipolar disorder, and severe anxiety disorders.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-08-17 (Actual); Study Completion 2025-09-17 (Actual)

PRIMARY OUTCOMES:
Assessment of sensory modulation scale (ASMS) | Baseline and 8 weeks
  The 141 items in the ASMS comprise 3 scales of 30, 30 and 21 items in these scales. First 30 items consist question of sensory over-responsive (SOR) and second 30 items consist questions of sensory under-responsive (SUR) and third 21 items consist questions of sensory seeking (SS) these all items use to evaluate children with mental, behavioural and neuro-developmental disorders, the cut of values of this questionnaire is given here. The participant will be given 1 score of each item if they answer "Yes" and will be given 2 score if they answer "No", the total score of 1ST & 2ND items SOR and SUR are 60. Minimum score, less than 30 show SOR and maximum score, greater than 30 show SUR and in 3rd item score less than 21 show SS.
Strength and difficulty questionnaire (SDQ) | Baseline and 8 weeks
  "Strengths and Difficulties" Parent and Teacher reported questionnaire for children aged 04-17 years is a behavioral measuring tool. The SDQ includes 25 items that examine a range of 'strengths and difficulties' as behavioral indicators of probable mental health disorders. The items contribute to 5 subscales, each with 5 items and a minimum score ranging from 0 (lowest score) to 10 (highest score): conduct difficulties, hyperactivity/inattention, emotional signs, problems with peers, and social conduct. The sum of the first 4 subscales yields a total difficulty score that ranges from 0 to 40

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Yousaf, MSPT(Peads), Principal Investigator — Riphah International University
Locations (1):
- Nishtar Medical University, Multan, Multan Khurd, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No